CLINICAL TRIAL: NCT06650280
Title: Assessment of Osseointegration of Dental Implants with Three Different Coatings for Early Loading Purpose and Marginal Bone Loss in the Posterior Maxilla. a Randomized Clinical Trial
Brief Title: Assessment of Rapid Osseointegration of Dental Implants with Different Coatings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Mahmoud Ismail, Lecturer of Oral & Maxillofacial Surgery, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31910-4
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Dental Implants; Hyaluronic Acid
Keywords: dental implants; rapid osseointegration; early loading
MeSH Terms: interventions — Hyaluronic Acid; nano-hydroxyapatite-collagen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- sandblasted acid etched group (Experimental): sandblasted acid etched coated implants will be allocated to this arm
  Interventions: Other: sandblasted acid etched
- nano-hydroxyapatite group (Active Comparator): nano-hydroxyapatite coated implants will be allocated to this arm
  Interventions: Other: nano-hydroxyapatite
- hyaluronic acid group (Experimental): hyaluronic acid coated implants will be allocated to this arm
  Interventions: Other: Hyaluronic Acid (HA)

INTERVENTIONS:
Other: Hyaluronic Acid (HA) — hyaluronic acid coated implants will be placed in posterior maxilla to evaluate rapid osseointegration
  Arms: hyaluronic acid group
Other: nano-hydroxyapatite — nano-hydroxyapatite coated implants will be placed in posterior maxilla to assess rapid osseointegration
  Arms: nano-hydroxyapatite group
Other: sandblasted acid etched — SLA coated implants will be placed in posterior maxilla and implant stability will be evaluated
  Arms: sandblasted acid etched group

SUMMARY:
The study will assess early osseointegration of dental implant with three different coating materials through secondary implant stability

DETAILED DESCRIPTION:
Dental implants with sandblasted acid itched coating, nano-hydroxyapatite coating, and hyalouronic acid coating will be placed in the posterior maxilla to restore a missing tooth. Implant stability by the use of Ostell will be measured immediately post-operative, 4, 6, and 12 weeks post-operative.

marginal bone loss around the implants will be compared immediately after final restoration delivery and after one year

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing at least one maxillary posterior tooth
2. Patients free from any systemic disease
3. Patients who approve to be included in the trial and sign the informed consent
4. Patients with no intra-bony defect.
5. Adults aged 18 years old and above

Exclusion Criteria:

1. Patients who are allergic to titanium
2. Heavy smoker patient
3. Patients receiving chemotherapy or radiotherapy
4. Patients who refused to be included in the trial

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
rapid osseintegration | immediately post-operative, 4, 6, and 12 weeks post-operative
  rapid osteointegration of dental implants will be evaluated by the use of Ostell device which measures primary and secondary stability expressed as ISQ measures ranging from zero till 90

SECONDARY OUTCOMES:
marginal bone loss | immediately after final restoration delivery and one year post-operative
  the bone height from implant's platform till implant's tip will be measured and compared between immediately after final restoration delivery and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamdy, Lecturer, Principal Investigator — Faculty of Dentistry, MSA University, Egypt
Locations (1):
- Faculty of Dentistry, MSA University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atsumi M, Park SH, Wang HL. Methods used to assess implant stability: current status. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):743-54. PMID 17974108